CLINICAL TRIAL: NCT00174525
Title: A Phase IIA, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose, Safety, Tolerability, Pharmacokinetic, Pharmacodynamic, and Immunogenicity Trial of AAB-001 in Patients With Mild to Moderate AD
Brief Title: Safety Study of Passive Immunization for Patients With Mild to Moderate Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pharmacology Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRI#585
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Caregivers; Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

INTERVENTIONS:
Drug: AAB-001

SUMMARY:
This research study will assess whether AAB-001 is safe, well tolerated and effective for use in patients with Alzheimer's Disease. AAB-001 is a new drug that is not available outside this study. AAB-001 is an antibody (a type of protein usually produced by white blood cells to destroy other substances in the body). In Alzheimer's disease a protein called amyloid gathers in the brain and is thought to cause symptoms like memory loss and confusion. It is hoped that AAB-001 will attach to the amyloid protein in your brain and help your body to remove it.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD
* Age from 50 to 85 years, inclusive
* Rosen Modified Hachinski ischemic score less than or equal to 4
* Magnetic Resonance Imaging (MRI) scan consistent with the diagnosis of AD
* Fluency in English
* Stable doses of medications

Exclusion Criteria:

* Significant neurological disease other than AD
* Major psychiatric disorder
* Significant systemic illness
* History of stroke or seizure
* Weight greater than 120kg (264 lbs.)
* History of autoimmune disease
* Smoking more than 20 cigarettes per day
* Anticonvulsants, anti-Parkinson's, anticoagulant, or narcotic medications
* Prior treatment with experimental immunotherapeutics or vaccines for AD
* Presence of pacemakers or foreign metal objects in the eyes, skin, or body

Ages: 50 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-04; Study Completion 2008-04

PRIMARY OUTCOMES:
Safety assessments

SECONDARY OUTCOMES:
Blood levels of administered study drug
Cognitive and functional assessments

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E. Grosz, MD, Principal Investigator — Pharmacology Research Institute, Northridge
Locations (2):
- United States (2):
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Northridge, California